CLINICAL TRIAL: NCT04042155
Title: Clinical Application Model of Direct Oral Anticoagulants (MACACOD). Comprehensive Management of ACOD From a Specialized Center in Antithrombotic Therapy and Its Area of Influence
Brief Title: Real-life Clinical Outcomes of Direct Oral Anticoagulants (MACACOD)
Acronym: MACACOD
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ACO-2018-31
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Recurrent Venous Thromboembolism
Keywords: dabigatran; rivaroxaban; apixaban; edoxaban
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism | interventions — Dabigatran; Rivaroxaban; apixaban; edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Plasma samples remaining from the routine blood tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: dabigatran, rivaroxaban, apixaban or edoxaban — Record of all serious complications associated with any of the drugs and the clinical changes that occurred during prospective follow-up.
  Other Names: Pradaxa, Xarelto, Eliquis or Lixiana

SUMMARY:
MACACOD is a clinical record in the usual clinical practice of direct oral anticoagulants (dabigatran, rivaroxaban, apixaban and edoxaban). Design: single-center, observational, prospective, uncontrolled study of anticoagulated patients with any direct oral anticoagulant (DOAC) with atrial fibrillation or venous thromboembolism to determine the incidence of serious complications (thromboembolic or hemorrhagic) in real life

DETAILED DESCRIPTION:
Population: Patients over 18 years of age, with recurrent atrial fibrillation or venous thromboembolism, already anticoagulated with any DOAC or patients who initiate therapy with DOAC and who give their consent. Upon entering the study, demographic data, previous anticoagulant treatments, previous serious complications, comorbidities and baseline analytical results are recorded. The risk scores CHA2DS2-Vasc, HAS-BLED and Charlson comorbidity index (CCI) are calculated. The type of health education received in relation to anticoagulant therapy is also recorded. During the follow-up, complications and clinical changes and the analytical results of coagulation, renal and hepatic function will be recorded. The risk scores will be updated at each visit. In case of serious complications, the associated costs will be estimated.

ELIGIBILITY:
Inclusion Criteria:

· Patients older than 18 years.

* With atrial fibrillation or recurrent venous thrombosis.
* In chronic treatment with any DOAC type drug.
* Patients who sign the informed consent

Exclusion Criteria:

* Patients who do not guarantee collaboration.
* Patients with advanced cognitive impairment and not supervised.
* Patients with alcoholism.
* Patients with psychiatric disorder and not supervised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under treatment with DOAC controlled at the Hospital de Sant Pau in Barcelona and in their area of influence (Primary Care Centers). These patients must be older than 18 years, with atrial fibrillation or recurrent venous thrombosis.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic events | 3 years
  Any documented embolic stroke, peripheral arterial embolism or venous thromboembolism
Major haemorrhagic events | 3 years
  Any documented bleeding event grade 3 or 5 in the Bleeding Assessment Research Consortium (BARC) scale Full scale name: Bleeding Assessment Research Consortium Scale ranges: 0-5 Where 0 is the better result and 5 is the worst

SECONDARY OUTCOMES:
Other thrombotic events | 3 years
  Myocardial infarction, transient ischemic attack, superficial thrombophlebitis
Clinically (non major) relevant bleeding | 3 years
  Any documented bleeding event grade 2 in the Bleeding Assessment Research Consortium (BARC) scale Full scale name: Bleeding Assessment Research Consortium Scale ranges: 0-5 Where 0 is the better result and 5 is the worst
Mortality | 3 years
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Souto, MD, PhD, Principal Investigator — Hospital de la Santa creu i Sant Pau - Barcelona
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No